CLINICAL TRIAL: NCT00510445
Title: A Phase I Study of GRN163L in Combination With Paclitaxel and Carboplatin in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of GRN163L With Paclitaxel and Carboplatin in Patients With Advanced or Metastatic Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRN163L CP14A005
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Lung Cancer
Keywords: Non Small Cell Lung Cancer; Advanced Non Small Cell Lung Cancer; Metastatic Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — imetelstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Trial (Experimental): Patients will be enrolled in the order of confirmation of eligibility. Dose cohorts will be filled sequentially with a minimum of 3 patients. Once assigned to a dose cohort, each patient will continue to be treated at the same dose level throughout the course of the study.
  Interventions: Drug: Imetelstat Sodium (GRN163L)

INTERVENTIONS:
Drug: Imetelstat Sodium (GRN163L) — The starting dose of GRN163L for this study will be 3.2 mg/kg. Subsequent dose levels will be 4.8, 6, 7.5, 9, 11, and 13.5 mg/kg. The maximum dose to be administered will not exceed 13.5 mg/kg.
  Paclitaxel and carboplatin will be administered on Day 2 of each 21-day cycle.

SUMMARY:
The purpose of this study is to determine the safety and the maximum tolerated dose (MTD) of GRN163L when administered in combination with a standard paclitaxel/carboplatin regimen to patients with advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
GRN163L is a telomerase template antagonist with in vitro and in vivo activity in a variety of tumor model systems. Telomerase is an enzyme that is active primarily in tumor cells and is crucial for the indefinite growth of tumor cells. Inhibition of telomerase may result in antineoplastic effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC
* Stage IIIb with pleural effusion, Stage IV, or recurrent disease
* Measurable or evaluable disease by RECIST criteria
* ECOG performance status 0-1
* Adequate hepatic/renal function and platelet count
* If previously treated with an anthracycline, anthracenedione, or trastuzumab, must have left ventricular ejection fraction > 50%

Exclusion Criteria:

* More than 2 prior chemotherapy regimens for metastatic disease (prior adjuvant chemotherapy is allowed)
* Tumor progression during treatment with paclitaxel (refractory to paclitaxel)
* Taxane-based regimen within 12 weeks
* Any systemic therapy for cancer within 4 weeks
* Anti-platelet therapy within 2 weeks, other than low dose aspirin prophylaxis therapy
* Therapeutic anticoagulation therapy except for low dose warfarin (eg, 1 mg by mouth per day)
* Radiation therapy within 3 weeks
* Major surgery within 4 weeks (central line placement is allowed)
* Prolongation of PT or aPTT > the ULN or fibrinogen < the LLN
* History of or active central nervous system metastatic disease
* Any other active malignancy
* Active or chronically recurrent bleeding (eg, active peptic ulcer disease)
* Clinically significant infection
* Active autoimmune disease requiring immunosuppressive therapy
* Clinically significant cardiovascular disease or condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety and MTD | First 3 weeks

SECONDARY OUTCOMES:
PK and efficacy | Baseline to end of treatment

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: Related Info — http://www.geron.com